CLINICAL TRIAL: NCT06861036
Title: Heterogeneity of Oral Squamous Cell Carcinoma Analysis by Single Cell RNA Sequencing
Acronym: HOASIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ET22-338 HOASIS
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Oral Squamous Cell Carcinomas
Keywords: scRNAseq; Heterogeneity of all cell population; OSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: A clinical-biological cohort of patients with OSCC.
  Samples:
  * 1 blood sample (6 mL)
  * 1 or 2 tumoral specimen (depending on the size of the tumor)
  * 1 specimen of the healthy oral mucosa
  * 1 leucoplakia specimen if applicable. The biospecimens will be collected at the time of the surgery scheduled in the standard routine medical care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinical-biological cohort (Other): A clinical-biological cohort of 50 patients with OSCC.
  Blood sample and biospecimen at the time of a standard surgery.
  Interventions: Procedure: Biospecimen; Procedure: Blood sampling

INTERVENTIONS:
Procedure: Biospecimen — * 1 or 2 tumoral specimen (depending on the size of the tumor)
  * 1 specimen of the healthy oral mucosa
  * 1 leucoplakia specimen if applicable.
  The biospecimens will be collected at the time of the surgery organised for the standard routine medical care.
Procedure: Blood sampling — Blood sampling (6 mL), taken from a routine biological exam.

SUMMARY:
The goal of this project is to characterise the heterogeneity of all cell populations (tumour cells, stromal and immune microenvironment) present in the tumor and their normal (and leucoplasic) counterparts by scRNAseq in OSCC patients.

DETAILED DESCRIPTION:
Epidermoid carcinomas of upper aerodigestive tract are the 8th most common cancers in the world. Worldwide, this represents more than 500.000 cases per year and 20.000 cases per year in France (statistics 2018-2020). Among these cancers, oral squamous cell carcinoma (OSCC) are the most common location, leading to significant morbidity and mortality.

OSCC treatment is based on surgery and/or radiotherapy and/or chemotherapy. Immune Check point Inhibitors (ICIs) targeting PD-1 have been approved for recurrent and metastasic OSCC. However, only 15-20% of these patients are treated thanks to this anti-PD-1. Thus, there is a real need to improve the efficacy of ICIs in the treatment of HNSCC. The scRNAseq is a method which allows to study the tumoral heterogeneity, the microenvironment and the dynamic and regulation mecanisms in cells cancer. This technology could improve patient stratification, identify pronostic biomarkers, constitute an important tool in the therapeutical take care and lead to understand tumoral evolution and develop new prevention strategies.

The aim of the study is to characterise the heterogeneity of all cell populations (tumour cells, stromal and immune microenvironment) present in the tumor and their normal (and leucoplasic) counterparts by scRNAseq in OSCC patients.

ELIGIBILITY:
Inclusion Criteria:

* I1. Male or female at least 18 years old.
* I2. Patient with OSCC and undergoing surgery at the Centre Léon Bérard.
* I3. Patient who has agreed to participate in this research and sign consent.
* I4. Patient affiliated to a medical insurance.

Exclusion Criteria:

* NI1. Pregnant or nursing woman.
* NI2. Contraindication to general anesthesia.
* NI3. Suspicion of rare tumor of particular histology other than squamous cell carcinoma (Sarcoma...).
* NI4. Patient under curatorial or guardianship or placed under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Characterization of the heterogeneity of all cell populations (tumour cells, stromal and immune microenvironment) present in the tumor and their normal (and leucoplasic) counterparts by scRNAseq in OSCC patients. | 3 years
  Transcriptomic data from scRNAseq for all cell populations

SECONDARY OUTCOMES:
Description of the functional interactions among tumor, stromal, and immune subpopulations identified by scRNAseq | 3 years
  Describe the functional interactions between tumor, stromal, and immune subpopulations using ex vivo culture models and co-culture assays. Cellular responses will be assessed using transcriptomic analysis and phenotypic characterization.
Correlation between refined patient stratification (based on tumor, stromal and immune sub-population) and the impact on the response to ex-vivo treatments. | 3 years
  Correlation between tumor, stromal and immune sub-populations likely to refine patient stratification and the impact on the response to ex-vivo treatments.
Identification of prognostic and predictive biomarkers for oral squamous cell carcinoma evolution | 3 years
  Correlation of gene expression profiles with disease progression to identify prognostic and predictive biomarkers in scRNAseq and bulk RNAseq datasets

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Zrounba, M.D., Principal Investigator — philippe.zrounba@lyon.unicancer.fr
Locations (1):
- Centre Léon Bérard, Lyon, France